CLINICAL TRIAL: NCT02334150
Title: Effects of Combined Spinal-epidural Analgesia During Labor on Postpartum Electrophysiological Function of Maternal Pelvic Floor Muscle: a Randomized Controlled Trial
Brief Title: Epidural Analgesia on Electrophysiological Function
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nanjing Maternity and Child Health Care Hospital (Other)
Responsible Party: Principal Investigator, Ji-Juan Xing, Nanning Maternity and Child Health Care Hospital, Nanjing Maternity and Child Health Care Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NanningMCH; Ji-Juan Xing (Registry Identifier: CSEAEF)
Record Dates: First submitted 2014-12-31; First posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Prolonged Labor; Healthy; Pelvic Floor Disorders
Keywords: combined spinal-epidural analgesia; pelvic floor muscle; postpartum electrophysiological function
MeSH Terms: conditions — Pelvic Floor Disorders | interventions — Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CSEA group (Experimental): Women in the CSEA group received CSEA during labor. An intravenous line was established when the uterine opening measured 1-2 cm. Then sufentanil (5-7 μg) was injected intrathecally. When the visual analogue pain score was 3 or higher, a mixture of ropivocaine (0.143%) and sufentanil (0.3 μg/ml) was continuously infused into the epidural space using an analgesia pump until the cervix was fully dilated. Load capacity was 5 ml. The analgesic plane was controlled under T10.
  Interventions: Drug: CSEA (ropivocaine and sufentanil)
- Control group (No Intervention): Women in the control group were not provided any analgesia during labor.

INTERVENTIONS:
Drug: CSEA (ropivocaine and sufentanil) — Women in the CSEA group received CSEA during labor. An intravenous line was established when the uterine opening measured 1-2 cm. Then sufentanil (5-7 μg) was injected intrathecally. When the visual analogue pain score was 3 or higher, a mixture of ropivocaine (0.143%) and sufentanil (0.3 μg/ml) was continuously infused into the epidural space using an analgesia pump until the cervix was fully dilated. Load capacity was 5 ml. The analgesic plane was controlled under T10.
  Other Names: Combined spinal-epidural analgesia
  Arms: CSEA group

SUMMARY:
Combined spinal-epidural analgesia (CSEA) is sometimes used for difficult births, but whether it contributes to postpartum pelvic muscle disorder is unclear. This randomized controlled trial examined whether CSEA affects the electrophysiological index of postpartum pelvic floor muscle during labor. The investigators plan to recruit 300 primiparous healthy women.

DETAILED DESCRIPTION:
Labor analgesia can relieve labor pain, reduce stress reactions, and improve blood supply to the fetus, benefiting mother and baby. Though traditional epidural analgesia has been used for more than 40 years, combined spinal-epidural analgesia (CSEA) has become popular because it provides faster-onset pain relief with minimal motor weakness. CSEA may also accelerate cervical dilation.

Despite the popularity of CSEA, whether it is associated with short- or long-term beneficial or adverse effects on mothers remains unclear. One question is whether the procedure affects the risk of female pelvic floor disorder (PFD), in which the pelvic floor muscles are injured. These muscles are responsible for supporting the pelvic organs and for stabilizing them during the rhythmic, strong labor contractions and for the diaphragm to contract enough to generate pressures of up to 19 kPa. Numerous risk factors have been associated with PFD, including obesity, diabetes, older age, connective tissue disorder, neurological disease, pregnancy, vaginal delivery and childbirth. PFD can lead in turn to stress urinary incontinence, overactive bladder, pelvic organ prolapse and fecal incontinence, all of which can strongly reduce women's physical and psychological health.

Pelvic floor function can be analyzed by measuring the strength and degree of fatigue of pelvic floor muscles, as well as the pelvic dynamic pressure. Abnormalities in these indicators appear even before patients complain of the signs and symptoms of PFD, making them a useful early diagnostic index.

In this randomized controlled study, we examined whether CSEA affects postpartum pelvic floor muscle function in primiparous mothers who give birth vaginally, as well as the duration of different stages of labor. Our results should help establish whether the widespread use of CSEA provides benefits to mothers or poses a risk.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women gave birth by vaginal delivery between June 2013 and June 2014 in the Maternal and Child Health Hospital of Nanning
* They were 22-30 years old
* They were 155-165 cm tall
* They were assigned a score of I or II on the American Society of Anesthesiologists scale
* They gave birth by vaginal delivery to a live, single, mature fetus (≥ 38, ≤ 40 w) in the head position
* A neonatal weight of 2900-3500 g

Exclusion Criteria:

* History of chronic cough
* Chronic constipation or pelvic organ resection
* Family history of urinary incontinence
* Pelvic organ prolapsus
* Any systemic disease before delivery
* A history of surgery, trauma, tumors or deformity of lumbar vertebrae

Ages: 22 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 308 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Muscle strength scores | 6 weeks
  The postpartum strength of pelvic floor muscles was measured with subjects in the supine lithotomy position. A vaginal manometric probe with a balloon was sheathed with a condom and placed into the vagina; the top of the device lay at the bottom of the vagina before air inflation. The other side of the probe was connected to the PHENIX muscle stimulator. Muscle strength was assessed using the international muscle strength detection method, which features a strength scale from 0 to 5. The strength score depends on whether vaginal muscle contraction upon stimulation fails to occur (0 points) or lasts 1 second (1 point), 2 seconds (2 points) and so on. If the contraction lasts 5 seconds or more, a strength score of 5 is assigned.

SECONDARY OUTCOMES:
Degrees of muscle fatigue | 6 weeks
  Degree of muscle fatigue was considered normal if 0%, abnormal if <0%.
The distribution of pelvic floor dynamic pressures | 6 weeks
  Pelvic floor dynamic pressure was considered normal when it fell between 80 and 150 cm H2O.

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Juan Xing, Principal Investigator — Maternal and Child Health Hospital of Nanning City
Locations (1):
- Maternal and Child Health Hospital of Nanning City, Nanning, Guangxi, China

REFERENCES:
- [Background] Frawley HC, Galea MP, Phillips BA, Sherburn M, Bo K. Effect of test position on pelvic floor muscle assessment. Int Urogynecol J Pelvic Floor Dysfunct. 2006 Jun;17(4):365-71. doi: 10.1007/s00192-005-0016-3. Epub 2005 Oct 5. PMID 16205845
- [Result] Caroci Ade S, Riesco ML, Sousa Wda S, Cotrim AC, Sena EM, Rocha NL, Fontes CN. Analysis of pelvic floor musculature function during pregnancy and postpartum: a cohort study: (a prospective cohort study to assess the PFMS by perineometry and digital vaginal palpation during pregnancy and following vaginal or caesarean childbirth). J Clin Nurs. 2010 Sep;19(17-18):2424-33. doi: 10.1111/j.1365-2702.2010.03289.x. PMID 20920070
- [Derived] Xing JJ, Liu XF, Xiong XM, Huang L, Lao CY, Yang M, Gao S, Huang QY, Yang W, Zhu YF, Zhang DH. Effects of Combined Spinal-Epidural Analgesia during Labor on Postpartum Electrophysiological Function of Maternal Pelvic Floor Muscle: A Randomized Controlled Trial. PLoS One. 2015 Sep 4;10(9):e0137267. doi: 10.1371/journal.pone.0137267. eCollection 2015. PMID 26340002